CLINICAL TRIAL: NCT02725775
Title: A Study of the Acute and Chronic Effects of 100% Florida Orange Juice Consumption on Cognitive Performance in 7-10 Year Old UK School Children
Brief Title: Acute and Chronic Effects of 100% Florida Orange Juice Consumption on Cognitive Performance in 7-10 Year Old Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leeds (Other)
Collaborators: Department of Citrus, State of Florida USA (Unknown); University of East Anglia (Other)
Responsible Party: Principal Investigator, Prof Louise Dye, Professor, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: RFP 15-01
Record Dates: First submitted 2016-03-22; First posted 2016-04-01 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Healthy
Keywords: Orange Juice, Polyphenol, Cognition

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 100% OJ (Active Comparator): 240ml 100% Florida Orange Juice consumed on a daily basis for 10 weeks.
  Interventions: Dietary Supplement: 100% Florida OJ
- Equicaloric Orange Drink (Placebo Comparator): An equicaloric placebo orange drink (containing equivalent dose of sucrose, glucose, fructose, vitamin C and citric acid for flavour) consumed daily for 10 weeks.
  Interventions: Dietary Supplement: Placebo Equicaloric Orange Drink

INTERVENTIONS:
Dietary Supplement: 100% Florida OJ
  Arms: 100% OJ
Dietary Supplement: Placebo Equicaloric Orange Drink
  Arms: Equicaloric Orange Drink

SUMMARY:
This study is a 10-week intervention study to examine the acute and chronic effects of daily intake of a 100 % orange juice drink vs control drink on cognitive performance. The study aims to determine if there are any benefits of whole orange juice intake on cognitive performance acutely (i.e. an improvement in performance at week 1) and chronically (i.e. an improvement in performance at week 10).

DETAILED DESCRIPTION:
This study will employ a randomised 10 week, parallel groups, double blind, placebo controlled design to investigate the effects of daily supplemental orange juice compared with an equicaloric placebo orange drink on cognitive performance in 7-10 year old school children. Following screening, participants will be randomly assigned to one of two conditions: (1) Active group: 100% orange juice, (2) Placebo group: control drink (containing equivalent dose of sucrose, glucose, fructose, vitamin C and citric acid for flavour). Both the active and control groups will receive a drink daily for 10 weeks delivered as a school-based morning intervention administered by researchers. Children will also be given drinks to consume over the weekends and school holidays monitored by a drink intake diary. Participants, parents and teachers will be blind to their assigned condition. Researchers will also be blinded until completion of the data analysis.

Following a practise session at screening (week -1) to familiarise the participants with the cognitive tests and study drinks, participants will take part in 3 test sessions - at baseline (Week 0), on Day 1 of intervention (start of Week 1; acute effects) and immediately post intervention (end of Week 10; chronic effects).

At week -1 (screening) children will be tested for colour blindness (Ishihara test) and complete the Wechsler abbreviated scale of intelligence (WASI) for screening purposes. Respiratory peak flow, height, and weight will also be measured to examine the relationship between cognitive performance and physical activity.

This study design, including both the test day and morning juice supplementation, is intended to emulate the children's normal routine as far as possible. Each carton of juice will be provided mid-morning to act as a supplement to their usual diet.

Measures:

The cognitive tests included in the study are listed below:

* Immediate and delayed picture recognition
* Delayed spatial memory
* Tower of Hanoi (executive function - planning/strategy)
* Corsi block tapping test (executive function and working memory)

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 7-10 years
* Willingness to consume test drinks during the study (determined by a score of 5 on the taste testing Likert scale for both orange juice drinks [attached])
* Ability to follow verbal and simple written instructions in English
* Ability to give written consent
* Normal vision, with appropriate corrective lenses if required
* Ability to understand cognitive testing instructions and responding requirements

Exclusion Criteria:

* Poor general health
* Colour blindness (to be assessed at screening using Tests for Colour Blindness (Isihara, 1951)
* Behavioural difficulties or attention disorders (e.g. Attention Deficit Hyperactivity Disorder)
* Learning disabilities which interfere with the ability to understand written or verbal communications
* Inability to understand the objective of the cognitive tests, or carry out the tests
* Any food allergies or intolerances to study drinks
* Acute illness, or feelings of unwell, within the week prior to testing
* Current administration of any psychotropic medication or supplementation in the month prior to testing, or during testing
* Hearing impairment that precludes the ability to follow verbal instructions

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2016-03; Primary Completion 2017-03 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Immediate and delayed picture recognition | Acute = 3 hours post first consumption. Chronic = After 10 weeks daily consumption
  Primary dependent variable: number of pictures successfully recalled (from 20 presented) immediately following presentation and after a delay consisting of two cognitive tests (Corsi Tapping and Tower of Hanoi).

SECONDARY OUTCOMES:
Delayed spatial memory | Acute = 3 hours post first consumption. Chronic = After 10 weeks daily consumption
  Primary dependent variable: number of spatial patterns successfully recognised from initial presentation (14 patterns presented twice). Recognition memory paradigm showing participants two patterns; one which was shown in the presentation phase and one which was not and requesting the participant select the presented pattern. Between presentation and recognition phases the participants engaged in a Corsi tapping test and a Tower of Hanoi test.
Tower of Hanoi (executive function) | Acute = 3 hours post first consumption. Chronic = After 10 weeks daily consumption
  Executive function - planning/strategy. Primary dependent variables: number of correctly solved puzzles and number of errors. Participants complete 2 trials at 8 levels of difficulty (difficulty indexed by number of moves required to complete the puzzle).
Corsi block tapping test (Executive function and working memory) | Acute = 3 hours post first consumption. Chronic = After 10 weeks daily consumption
  Executive function and working memory. Primary dependent variables: number of correctly recalled "block" presentations. An array of 9 white boxes are presented. Individual boxes are illuminated in sequences of increasing number of target presentations (2 - 8 boxes illuminated). After each pattern sequence is completed, participants are presented with the blank array of white boxes and are required to repeat the pattern in sequential order.

CONTACTS AND LOCATIONS:
Overall Officials: Clare Lawton, PhD, Principal Investigator — University of Leeds
Locations (1):
- Human Appetite Research Unit, University of Leeds, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided